CLINICAL TRIAL: NCT04273100
Title: PD-1 mAb Combined With Lenvatinib and TACE in the Treatment of BCLC B/C Hepatocellular Carcinoma: Single Arm, Single Center, Non Randomized, Open Label Study
Brief Title: PD-1 Monoclonal Antibody, Lenvatinib and TACE in the Treatment of HCC
Acronym: PLTHCC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PLTHCC
Record Dates: First submitted 2020-01-28; First posted 2020-02-17 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-01

CONDITIONS: Hepatocellular Carcinoma Non-resectable
Keywords: Hepatocellular carcinoma; Immune Suppression; Angiogenesis; Hepatic Artery Embolism
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — lenvatinib

STUDY DESIGN:
Intervention Model Description: This study focuses on the in-operable, middle and late stage (BCLC-B and BCLC-C) HCC patients. The participants will receive the combined treatment of immunotherapy (PD-1 monoclonal antibody), local therapy (TACE) and anti-angiogenic therapy (lenvatinib).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): The participants will receive the combined treatment of immunotherapy (PD-1 monoclonal antibody), local therapy (TACE, lobaplatin and epirubicin and anti-angiogenic therapy (lenvatinib)
  Interventions: Combination Product: PD-1 mAb combined with TACE and lenvatinib

INTERVENTIONS:
Combination Product: PD-1 mAb combined with TACE and lenvatinib — the combination of immunotherapy (PD-1 monoclonal antibody), local therapy (TACE) and anti-angiogenic therapy (lenvatinib)

SUMMARY:
The vast majority of primary liver cancer (90%) is hepatocellular carcinoma (HCC), and the majority of HCC patients have been locally advanced or metastatic disease when they are diagnosed in clinics. Most of them are not suitable for radical treatment. In the case of supportive treatment, the median survival time was only 7.9 months. Therefore, there is an urgent need for effective treatment for these patients.

At present, the overall objective response rate (ORR) of single or sequential therapy is not satisfied, and the over survival (OS) improvement is not ideal. Therefore, combined therapy maybe the good choice for patients with advanced HCC.

This study focuses on the in-operable, middle and late stage (BCLC-B and BCLC-C) HCC patients. Through the combination of immunotherapy (PD-1 monoclonal antibody), local therapy (TACE) and anti-angiogenic therapy (lenvatinib), it is expected to change the tumor microenvironment, restore the immune response, strengthen the anti-tumor effect of various treatments, and improve the therapeutic efficacy in patients with middle and late stage HCC.

DETAILED DESCRIPTION:
This study is a single arm, single center, non randomized, open label study. It is estimated that 56 patients with advanced HCC who can not receive radical resection will be enrolled.

The trial period of subjects includes screening period, treatment period and follow-up period.

The drug treatment was 240 mg of PD-1 monoclonal antibody, intravenous infusion on the first day, every 21 days as a treatment cycle; lenvatinib mesylate capsule, 12 mg (body weight ≥ 60 kg) or 8 mg (body weight < 60 kg), oral once a day, continuous oral; TACE, the blank microspheres and lobaplatin (30 mg) + epirubicin (40 mg) were injected into the hepatic artery by routine procedure, repeated every 4-6 weeks, and administered for 2-4 cycles. Treatment continues until the disease progresses, intolerable toxicity occurs, new anti-tumor treatment is started, informed consent is withdrawn, follow-up is lost, death occurs or treatment termination is required。

Screening will be performed between days - 21 and - 4. Informed consent was signed up to 4 weeks prior to the first day of cycle 1 before any screening procedure or evaluation was performed and the trial was fully explained to each subject.

Baseline evaluation results must be collected prior to the first trial drug administration (day 1 of cycle 1). Baseline assessments may be performed between days - 3 and - 1 or on day 1 of cycle 1. If performed within 3 days before the first day of cycle 1, the screening results can be used as baseline results.

The tumor imaging was evaluated every 8 weeks (± 7 days) since the first administration, and every 12 weeks (± 7 days) after 36 weeks. If there are clinical indications for disease progression, tumor evaluation is more frequent. In the event of disease progression, unacceptable toxicity, the subject's request to discontinue the trial or the subject's withdrawal of consent, the subject will discontinue the trial treatment.

When the trial treatment is stopped, the treatment visit shall be stopped within 7 days after the treatment is stopped in order to stop the treatment examination.

After the end of the treatment period (up to 2 years), subjects who can benefit from the study drug will continue to study the treatment of the drug until disease progression, intolerable adverse reactions, withdrawal of intensive care facility (ICF), other anti-tumor treatment, loss of follow-up, death or termination of the study.

After the occurrence of a clinical event, if it is judged by the investigators that it should be attributed to the progress of the disease and it is unlikely to recover even if the patient continues to receive treatment, it can be evaluated as clinical deterioration. It is up to the investigator to discuss and decide whether to continue or stop the treatment for the subject and record in the study file.

At the end of the study, subjects who are still under study treatment can continue to receive treatment through another extended study or other forms at the discretion of the investigator if they are stable or relieved in the efficacy evaluation and can tolerate the adverse reactions.

ELIGIBILITY:
Inclusion Criteria:

1. HCC confirmed by histology / cytology.
2. Age ≥ 18 years old.
3. Eastern Cooperative Oncology Group (ECOG) physical state score 0 or 1.
4. Barcelona clinical liver cancer (BCLC) stage B or stage C.
5. Participants who have not received other systemic anti-tumor treatment for HCC before the first administration, or who have received treatment but PD or SD ≥ 4 weeks.
6. Patients who had not received TACE before the first administration, or who had received TACE but SD ≥ 4 weeks.
7. According to RECIST v1.1, there is at least one measurable lesion.
8. Child Pugh score ≤ 7.
9. Participant has sufficient organ and marrow functions.
10. Expected survival time ≥ 12 weeks.
11. For women of childbearing age or male patients whose sexual partners are women of childbearing age, effective contraceptive measures should be taken during the whole treatment period and 6 months after the last medication.
12. Sign the written informed consent, and be able to follow the visit and relevant procedures specified in the plan

Exclusion Criteria:

1. Fibrolamellar carcinoma, sarcomatoid carcinoma, cholangiocarcinoma and other components previously confirmed by histology / cytology.
2. History of hepatic encephalopathy or liver transplantation.
3. Pleural effusion, ascites and pericardial effusion with clinical symptoms requiring drainage.
4. Acute or chronic active hepatitis B or C infection, hepatitis B virus (HBV-DNA) > 10^6 copies / ml; hepatitis C virus (HCV-RNA) > 10^3 copies / ml; HBsAg and anti HCV antibody were positive at the same time.
5. There is central nervous system metastasis.
6. Bleeding of esophageal or gastric varices caused by portal hypertension occurred in the past 6 months, or severe (G3) varices were found in endoscopic examination within 3 months before the first administration, or evidence of portal hypertension (including splenomegaly found in imaging examination) was found. The researchers assessed that the risk of bleeding was high and did not receive sclerotherapy or ligation under the endoscope.
7. The previous 6-month history of arteriovenous thromboembolism, including myocardial infarction, unstable angina, cerebrovascular accident, pulmonary embolism, deep vein thrombosis or any other serious thromboembolism. The thrombus of implanted vein port or catheter source or superficial vein is stable after routine anticoagulant treatment. Prophylactic use of low-molecular-weight heparin (e.g., enoxaparin 40 mg / day) is permitted.
8. Tumor thrombus of main portal vein, or involving superior mesenteric vein at the same time.
9. Aspirin (> 325 mg / day) or other drugs known to inhibit platelet function such as dipyridamole or clopidogrel were used for 7 consecutive days within 2 weeks before the first administration.
10. For uncontrolled hypertension, systolic blood pressure > 150 mmHg or diastolic blood pressure > 100 mmHg after the best medical treatment, hypertension crisis or hypertension encephalopathy history.
11. Symptomatic congestive heart failure (New York Heart Association class II-IV). Symptomatic or poorly controlled arrhythmias. The corrected QT interval (QTc) for the history or screening of congenital long QT syndrome was more than 500 ms (calculated by Fridericia method).
12. Serious bleeding tendency or coagulation dysfunction, or undergoing thrombolysis.
13. In the past 6 months, there was a history of gastrointestinal perforation and / or fistula, a history of intestinal obstruction (including incomplete intestinal obstruction requiring parenteral nutrition), extensive enterotomy (partial colectomy or extensive enterotomy with chronic diarrhea), Crohn's disease, ulcerative colitis or long-term chronic diarrhea.
14. Received radiotherapy within 3 weeks before the first administration. For patients who received radiotherapy three weeks before the first administration, all the following conditions must be met before entering the group: at present, there is no toxic reaction related to radiotherapy, no need to take glucocorticoids, excluding radiation pneumonia, radiation hepatitis, radiation enteritis, etc.
15. Previous and current pulmonary fibrosis history, interstitial pneumonia, pneumoconiosis, drug-related pneumonia, severe impairment of lung function and other lung diseases.
16. Active tuberculosis (TB), who is receiving anti TB treatment or has received anti TB treatment within one year before the first administration.
17. People with HIV infection (HIV 1 / 2 antibody positive) and known syphilis infection. Serious infection in active stage or poor clinical control.
18. Severe infection within 4 weeks before the first administration, including but not limited to hospitalization due to complications of infection, bacteremia or severe pneumonia.
19. Active autoimmune diseases requiring systemic treatment (such as the use of disease alleviation drugs, corticosteroids or immunosuppressants) occurred within 2 years before the first administration. Alternative therapies (e.g. thyroxine, insulin, or physiological corticosteroids for adrenal or pituitary insufficiency) are permitted. Known history of primary immunodeficiency. Only the patients with positive autoimmune antibody need to confirm whether there is autoimmune disease according to the judgment of researchers.
20. Immunosuppressive drugs were used within 4 weeks before the first administration, excluding local glucocorticoids or systemic glucocorticoids (i.e. no more than 10 Mg / day prednisone or the equivalent dose of other glucocorticoids), allowing temporary use of glucocorticoids due to dyspnea symptoms in the treatment of asthma, chronic obstructive pulmonary disease and other diseases.
21. Receive live attenuated vaccine within 4 weeks before the first administration or during the study period.
22. Major surgical procedures (craniotomy, thoracotomy or open hand) were performed within 4 weeks before the first administration (surgery) or an unhealed wound, ulcer, or fracture.
23. Received local treatment for liver cancer within 4 weeks before the first administration.
24. Chinese medicine with anti-tumor indications or drugs with immunomodulatory effects (including thymosin, interferon, interleukin, except for local use for control of pleural fluid or ascites) were received within 2 weeks before the first administration.
25. Uncontrolled / uncorrectable metabolic disorder or other non malignant organ disease or systemic disease or cancer secondary reaction, which may lead to higher medical risk and / or uncertainty of survival evaluation.
26. Known to be allergic to any PD-1 monoclonal antibody component.
27. Women of childbearing age who are unwilling or unable to use acceptable methods of contraception during the whole treatment period of this trial and within 12 weeks after the last administration of the study drug (women of childbearing age include: any women who have had menarche, and have not undergone successful artificial sterilization (hysterectomy, bilateral tubal ligation, or bilateral ovariectomy), pregnancy or lactation Women; women with positive pregnancy test results at the time of inclusion or before study drug administration; If the partner is a woman of childbearing age, the subject is a fertile male without effective contraceptive measures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2019-11-14 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
objective response rate (ORR) | Change from baseline tumor volume at 6 month
  The proportion of patients whose tumor volume reduction reaches the predetermined value and can maintain the minimum time limit. It is the sum of the proportion of complete response (CR) and partial response(PR). That is, ORR = CR + PR

SECONDARY OUTCOMES:
progression free survival (PFS) | Up to 24 months, from date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  Progression free survival period refers to the period from the beginning of treatment to the time when patients with cancer progress is observed or death occurs for any reason.
time to progression (TTP) | Up to 24 months, from date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  Time from the beginning of treatment to the objective progression of tumor
disease control rate (DCR) | 1 year
  It is the sum of the proportion of complete response (CR), partial response(PR) and stable disease(SD). That is, DCR = CR + PR + SD
duration of response | up to 48 weeks
  the time from the first evaluation of the tumor as CR or PR to the first evaluation as PD or any cause of death
overall survival | 1 year
  the time from the beginning of treatment to death caused by any reason (the last follow-up time is for the patients who lost the visit; the end of the study is for the patients who are still alive)

OTHER OUTCOMES:
conversion rate of hepatectomy | 1 year
  The ratio of patients with locally advanced liver cancer who could not be operated on before to get radical operation through comprehensive treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Hospital, Tianjin, Tianjin Municipality, China